CLINICAL TRIAL: NCT03565640
Title: Randomized Trial Comparing Anchorsure® Suture Anchoring System and the CapioTM Slim Suture Capturing Device for Sacrospinous Ligament Suspension.
Brief Title: Anchorsure Versus Capio for Sacrospinous Ligament Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00051211
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: Buttock pain; Thigh pain; Sacrospinous ligament fixation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants and research staff will be masked during the study as much as possible, however there will be a description of the type of sacrospinous ligament fixation device used within the body of the operative note for each patient that research staff could gain access to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Capio Slim Device (Active Comparator): Participants will be randomized to the sacrospinous ligament fixation with use of Capio Slim Device
  Interventions: Device: Capio Slim Device
- Anchorsure Device (Experimental): Participants will be randomized to the sacrospinous ligament fixation with use of Anchorsure Device
  Interventions: Device: Anchorsure Device

INTERVENTIONS:
Device: Capio Slim Device — Participants who have been assigned to sacrospinous ligament fixation for pelvic organ prolapse will have sacrospinous ligament fixation performed with the Capio Slim Device.
  Arms: Capio Slim Device
Device: Anchorsure Device — Participants who have been assigned to sacrospinous ligament fixation for pelvic organ prolapse will have sacrospinous ligament fixation performed with the Anchorsure Device.
  Arms: Anchorsure Device

SUMMARY:
Sacrospinous ligament fixation is a common method of repairing apical support for pelvic organ prolapse but it currently suffers from a high rate of postoperative buttock and posterior thigh pain. Anchorsure® is a relatively new FDA-approved device that uses an anchor instead of the widely-used suture capturing mechanism to perform sacrospinous ligament fixation. The study hypothesis is that Anchorsure® will reduce the degree and rate of buttock and posterior thigh pain compared to the widely used Capio™ Slim suturing capturing Device.

DETAILED DESCRIPTION:
Sacrospinous ligament fixation is a common method of repairing apical support for pelvic organ prolapse but it currently suffers from a high rate of postoperative buttock and posterior thigh pain. Rates of buttock and thigh pain 6 weeks after sacrospinous ligament fixation with the widely used Capio™ Slim device (Boston Scientific) are about 15-16% with immediate postoperative pain occurring in 55-84% of patients. This study is a randomized controlled single-blind study with the primary goal of investigating if there is an improvement in the intensity and rate of buttock and posterior thigh pain 1 day, 7 days, 6 weeks, and minimum 12 months after sacrospinous ligament fixation with a new device, the Anchorsure® Suture Anchoring System (Neomedic) compared to the widely utilized Capio™ Slim (Boston Scientific) device. 60 patients will be enrolled to undergo sacrospinous ligament fixation for treatment of pelvic organ prolapse. The patients will be randomized into two study groups; one will have sacrospinous ligament fixation using the Capio™ Slim device and the other with the Anchorsure® device. The patient's pain will be recorded via the numerical rating scale (NRS), a validated pain evaluation tool. The study is powered to detect a 2.5 point difference in pain between the two groups, a value that has been shown in studies to be clinically significant to acute pain patients. Secondary outcomes of surgeon satisfaction and efficiency with the devices will be assessed via surgeon questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* At least 21 years of age
* Surgical plan that includes a native tissue vaginal repair with apical support via sacrospinous ligament fixation. We will permit both hysteropexy and post-hysterectomy sacrospinous ligament suspension
* Understanding and acceptance of the need to return for the 6 week follow-up visit
* English speaking and able to give informed consent
* Willing and able to complete all study questionnaires
* Ambulatory

Exclusion Criteria:

* Prior sacrospinous ligament fixation procedure.
* Any serious disease or chronic condition that could interfere with the study compliance
* Inability to give informed consent
* Pregnancy or planning pregnancy prior to the 6 week postoperative visit
* Prior pelvic radiation
* Incarcerated
* Prior augmented (synthetic mesh, autologous graft, xenograft, allograft) prolapse repair
* History of significant buttock or leg pain in the past 3 months
* History of fibromyalgia, polymyositis, dermatomyositis, systemic lupus erythematosus, or other auto-immune myalgic conditions
* Current regular opioid drug therapy for any chronic pain condition
* History of loss of motor or sensory function of the lower extremities
* History of sacral decubitus ulcers
* Planned concomitant levatorplasty; anal sphincteroplasty, anal fissurectomy, rectopexy, or hemorrhoidectomy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have biological female reproductive organs.
Enrollment: 48 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data from the study will be kept on password protected digital storage for at least three years following the project completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At least 3 years from study completion
Access Criteria: Contact the principal investigator Dr. Catherine Matthews

REFERENCES:
- [Background] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- [Background] Atherton MJ, Daborn JP, Tsokos N, Jeffery JT, Yin MJ. Complications associated with tissue anchor migration after vaginal surgery using the tissue fixation system - a case series. Aust N Z J Obstet Gynaecol. 2012 Feb;52(1):83-6. doi: 10.1111/j.1479-828X.2011.01383.x. Epub 2011 Dec 6. PMID 22141331
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Brennand EA, Bhayana D, Tang S, Birch C, Murphy M, Cenaiko D, Ross S, Robert M. Anchor placement and subsequent movement in a mesh kit with self-fixating tips: 6-month follow-up of a prospective cohort. BJOG. 2014 Apr;121(5):634-40. doi: 10.1111/1471-0528.12536. Epub 2014 Jan 13. PMID 24621073
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Cepeda MS, Africano JM, Polo R, Alcala R, Carr DB. What decline in pain intensity is meaningful to patients with acute pain? Pain. 2003 Sep;105(1-2):151-7. doi: 10.1016/s0304-3959(03)00176-3. PMID 14499431
- [Background] DeLancey JO. Anatomic aspects of vaginal eversion after hysterectomy. Am J Obstet Gynecol. 1992 Jun;166(6 Pt 1):1717-24; discussion 1724-8. doi: 10.1016/0002-9378(92)91562-o. PMID 1615980
- [Background] Eilber KS, Alperin M, Khan A, Wu N, Pashos CL, Clemens JQ, Anger JT. Outcomes of vaginal prolapse surgery among female Medicare beneficiaries: the role of apical support. Obstet Gynecol. 2013 Nov;122(5):981-987. doi: 10.1097/AOG.0b013e3182a8a5e4. PMID 24104778
- [Background] Farrar JT, Berlin JA, Strom BL. Clinically important changes in acute pain outcome measures: a validation study. J Pain Symptom Manage. 2003 May;25(5):406-11. doi: 10.1016/s0885-3924(03)00162-3. PMID 12727037
- [Background] Ferrando CA, Walters MD. A randomized double-blind placebo-controlled trial on the effect of local analgesia on postoperative gluteal pain in patients undergoing sacrospinous ligament colpopexy. Am J Obstet Gynecol. 2018 Jun;218(6):599.e1-599.e8. doi: 10.1016/j.ajog.2018.03.033. Epub 2018 Mar 31. PMID 29614274
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Hsu Y, Chen L, Summers A, Ashton-Miller JA, DeLancey JO. Anterior vaginal wall length and degree of anterior compartment prolapse seen on dynamic MRI. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jan;19(1):137-42. doi: 10.1007/s00192-007-0405-x. Epub 2007 Jun 20. PMID 17579801
- [Background] Inoue H, Sekiguchi Y, Kohata Y, Satono Y, Hishikawa K, Tominaga T, Oobayashi M. Tissue fixation system (TFS) to repair uterovaginal prolapse with uterine preservation: a preliminary report on perioperative complications and safety. J Obstet Gynaecol Res. 2009 Apr;35(2):346-53. doi: 10.1111/j.1447-0756.2008.00947.x. PMID 19708181
- [Background] Karacaoglu MU, Ozyurek ES, Mutlu S, Odacilar E. Unilateral sacrospinous ligament fixation (USLF) with a mesh stabilizing anchor set: clinical outcome and impact on quality of life. Clin Exp Obstet Gynecol. 2016;43(2):216-9. PMID 27132413
- [Background] Maher CF, Murray CJ, Carey MP, Dwyer PL, Ugoni AM. Iliococcygeus or sacrospinous fixation for vaginal vault prolapse. Obstet Gynecol. 2001 Jul;98(1):40-4. doi: 10.1016/s0029-7844(01)01378-3. PMID 11430954
- [Background] Mowat A, Wong V, Goh J, Krause H, Pelecanos A, Higgs P. A descriptive study on the efficacy and complications of the Capio (Boston Scientific) suturing device for sacrospinous ligament fixation. Aust N Z J Obstet Gynaecol. 2018 Feb;58(1):119-124. doi: 10.1111/ajo.12720. Epub 2017 Sep 22. PMID 28940223
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Stanford EJ, Moore RD, Roovers JP, Courtieu C, Lukban JC, Bataller E, Liedl B, Sutherland SE. Elevate anterior/apical: 12-month data showing safety and efficacy in surgical treatment of pelvic organ prolapse. Female Pelvic Med Reconstr Surg. 2013 Mar-Apr;19(2):79-83. doi: 10.1097/SPV.0b013e318278cc29. PMID 23442504
- [Background] Summers A, Winkel LA, Hussain HK, DeLancey JO. The relationship between anterior and apical compartment support. Am J Obstet Gynecol. 2006 May;194(5):1438-43. doi: 10.1016/j.ajog.2006.01.057. Epub 2006 Mar 30. PMID 16579933
- [Background] Unger CA, Walters MD. Gluteal and posterior thigh pain in the postoperative period and the need for intervention after sacrospinous ligament colpopexy. Female Pelvic Med Reconstr Surg. 2014 Jul-Aug;20(4):208-11. doi: 10.1097/SPV.0000000000000091. PMID 24978086
- [Derived] Plair A, Smith W, Hines K, Schachar J, Parker-Autry C, Matthews C. Gluteal and Posterior Thigh Pain From a Suture Compared With an Anchor-Based Device in Patients Undergoing Sacrospinous Ligament Fixation: A Randomized Controlled Trial. Obstet Gynecol. 2022 Jan 1;139(1):97-106. doi: 10.1097/AOG.0000000000004629. PMID 34856573
- See also: FDA 2011 Urogynecologic Surgical Mesh: Update on the Safety and Effectiveness of Transvaginal Placement for Pelvic Organ Prolapse — https://www.fda.gov/downloads/medicaldevices/safety/alertsandnotices/UCM262760.pdf
- See also: SOUSA A, FLORES J, LEON J, SOUSA-GONZALEZ D. ICS 2017 Annual Meeting, Florence. Non-Discussion Video #850: RESULTS OF EFFICIENCY AND SAFETY IN REPAIRING PREVIOUS PROLAPSE THROUGH THE SURELIFT® SYSTEM. 5 YEARS RESULTS — https://www.ics.org/2017/abstract/850
- See also: AMAT L, GOMEZ A, MARTINEZ E, KAPLAN E. ICS 2010 Annual Meeting, Toronto. Non-Discussion Video #864: EVALUATION OF THE SAFETY AND EFFICACY OF PELVIC ORGAN PROLAPSE REPAIR USING SURELIFT® SYSTEM - PRELIMINARY RESULTS — https://www.ics.org/2010/abstract/864
- See also: Salicrú S. 2018 IUGA Annual Meeting, Vienna. Unmoderated Poster #503: Surgical repair of severe prolapse with Surelift System — https://iugameeting.org/program/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capio Slim Device | Anchorsure Device
Started | 23 | 24
Completed | 22 | 21
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capio Slim Device | Anchorsure Device | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (10.7) | 68.7 (8.8) | 69.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 19 | 38
  Black | 3 | 2 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (6.4) | 29.9 (6.6) | 30.0 (6.4)
POP-Q Stage Score [Mean (Standard Deviation); unit: Units on a scale] — The POP-Q assessment tool measures nine points in the vagina. The measurements are taken when woman is in the dorsal lithotomy position. The stages are: 0 if there is no prolapse at all, 1 if there is prolapse but the leading point is not within 1cm of hymen, 2 if the leading point is within 1 cm of hymen (from 1cm within the hymen to 1cm beyond the hymen), 3 if leading point is more than 1cm from the hymen but less than 2cm from being completely prolapsed, and 4 if leading point is within 2cm of being complete prolapsed. Higher POP-Q stages correlate to a worse degree of prolapse.
  Units on a scale | 2.7 (0.6) | 2.8 (0.8) | 2.7 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Buttock and Posterior Thigh Pain
Description: This will be assessed using the numeric rating scale (NRS). The score is 0-10, with higher scores denoting a greater degree of pain.
Time Frame: postoperative 12 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capio Slim Device | Anchorsure Device
Number analyzed (Participants) | 22 | 21
score on a scale
  Sacrospinous ligament fixation site Pain compared to preop | -0.5 (1.6) | -0.2 (0.9)
  Worst pain compared to preop | -1.8 (3.1) | -1.5 (2.8)

2. Secondary Outcome: POP-Q Stage Score
Description: The stage is assigned as follows: 0 if there is no prolapse at all, 1 if there is prolapse but the leading point is not within 1cm of the hymen, 2 if the leading point is within 1 cm of the hymen (from 1cm within the hymen to 1cm beyond the hymen), 3 if the leading point is more than 1cm from the hymen but less than 2cm from being completely prolapsed, and 4 if the leading point is within 2cm of being complete prolapsed. Therefore higher POP-Q stages correlate to a worse degree of prolapse than lower POP-Q stages.
Time Frame: at 12 MONTHS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Capio Slim Device | Anchorsure Device
Number analyzed (Participants) | 18 | 19
Units on a scale | 0.8 (0.9) | 0.9 (0.8)

3. Secondary Outcome: Change in Pelvic Flore Disability Index - 20 (PFDI-20) Scores From Baseline to 12 Months
Description: Symptomatic success was assessed by the pelvic floor disability index (PFDI-20) questionnaire. The PFDI-20 has 20 items within 3 sub-scales of symptoms (total of 20 items). Each item produces a response of 0 to 4, the average response in each sub-scale is multiplied by 25 to obtain the sub-scale score (range 0 to 100). The total score is the sum of the three sub-scale scores with a range of 0-300. Higher value for a time-point score indicates a greater degree of symptom bother.
  The difference in scores across the study time-points was calculated by subtracting the total score at baseline from the score at 12 months post-operation. A negative value for the difference in scores from baseline to 12 months indicates symptom improvement, where the more negative the difference in score is the greater the improvement in symptoms.
Time Frame: Baseline and Month 12
Population: These are the two study groups where patients were randomized to either have the Anchorsure or Capio Slim device used for their sacrospinous ligament fixation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capio Slim Device | Anchorsure Device
Number analyzed (Participants) | 22 | 21
score on a scale | -66.3 (64.4) | -71.0 (45.5)

4. Secondary Outcome: Change in Symptomatic Success - PFIQ-7 Scores
Description: Symptomatic success will be assessed by the Pelvic Floor Impact Questionnaire - 7 (PFIQ-7). The PFIQ-7 has 7 items for each of 3 sub-scales (total of 21 items). Each item produces a response of 0 to 3, the average response in each sub-scale is multiplied by 100/3 to obtain the total scale score (range 0 to 100). The total score is the sum of the three sub-scale scores with a range of 0-300. Higher value for a time-point score indicates a greater degree of symptom bother.
  The difference in scores across the study time-points was calculated by subtracting the total score at baseline from the score at 12 months post-operation. A negative value for the difference in scores from baseline to 12 months indicates symptom improvement, where the more negative the difference in score is the greater the improvement in symptoms.
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capio Slim Device | Anchorsure Device
Number analyzed (Participants) | 22 | 21
score on a scale | -26.4 (65.7) | -40.6 (62.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for an average of 15.4 months with standard deviation of (4.3). This is based on patient's time to approximately 1 year follow-up
Arm/Group | Capio Slim Device | Anchorsure Device
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03565640/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03565640/ICF_001.pdf